CLINICAL TRIAL: NCT07262385
Title: Calmer Brains: A Pilot Randomized Trial to Explore Structural and Functional Brain Development in Preterm Infants
Brief Title: Calmer Brains in Very Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Manon Ranger, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H25-01015
Record Dates: First submitted 2025-07-04; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Premature Infant
Keywords: Prematurity; Brain development; Stress; NICU; Pilot RCT; Feasibility; Calmer - therapeutic medical device
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: We will conduct a single-site, single-blind, two-group (treatment and control), randomized pilot trial and determine the feasibility of our study design. We will also gather preliminary data of Calmer's effect on infant structural and functional brain development to inform a larger trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calmer (Experimental): Infants in the Calmer group will have a Calmer* placed and left in their incubators for a minimum of 2 and maximum of 3 weeks and will receive treatment for a minimum cumulative total of 3 hours/day (i.e. time can be discontinuous).
  Each day, after the infant's parent rests for 10 minutes, the research and/or bedside nurse will record the heart and respiratory rates for a 2-minute period (or taken by the caregiver themselves after training by research/NICU staff). The 1-minute average will be used to program Calmer for each infant that day to better simulate day-to-day changes in infant-parent contact. The values can be adjusted over the day as parents wish.
  *Calmer, a patented, therapeutic bed that mimics key aspects of skin-to-skin care (SSC) to reduce stress in preterm infants. Calmer fits into NICU incubators and delivers 3 key SSC stimuli: touch, breathing motion, and heartbeat sounds (rates individualized to each infant based on their parents' HR/RR).
  Interventions: Device: Calmer
- Control (No Intervention): Infants in the Control group will receive standard NICU care, including parent SSC.

INTERVENTIONS:
Device: Calmer — Calmer, a unique, patented, therapeutic bed that mimics key aspects of SSC that reduce stress in preterm infants. Calmer fits into NICU incubators and cribs, and delivers 3 key SSC stimuli: touch, breathing motion, and heartbeat sounds; the rates of the latter 2 stimuli are individualized to each infant based on their parents' breathing and heart rates. Calmer is designed to provide complementary care only when parents are not able to give SSC. It is not meant nor designed to replace human SSC, so will never be tested as such a replacement. Instead, Calmer was invented to enhance and optimize brain development in preterm infants by reducing stress during the NICU stay, when parents/caregivers are not available for SSC. Our ultimate goal is to enable use of Calmer from an infant's admission to discharge, only during those times when caregivers are not available.
  Arms: Calmer

SUMMARY:
Very preterm infants in the neonatal intensive care unit (NICU) need lifesaving medical procedures which can be stressful and affect brain development. Calmer was invented to mimic key parts of parental holding (touch, heartbeat sounds and breathing motion) to help reduce stress if parents cannot be there to hold their infant. Using specialized brain scans done at full term, we will gather initial information in 22 infants born 3-4 months early to compare brain development in infants who receive Calmer at least 3 hours each day (+ regular NICU care) over 2-3 weeks with infants who have regular NICU care.

DETAILED DESCRIPTION:
Very preterm infants (< 32 weeks gestational age [GA]) experience developmentally unexpected, repeated stress as part of lifesaving care in the NICU during a period of considerable brain maturation and growth. Exposure to early-life stress alters brain maturation resulting in long-term changes in neurodevelopment. Parental skin-to-skin care (SSC) can mitigate stress; however, parents are not always available. Calmer, a patented, therapeutic medical device, was invented to simulate aspects of SSC (skin-like surface, breathing motion, heartbeat sounds) with rates of the latter two individualized for each infant. In a randomized trial, Calmer has been shown to stabilize brain blood flow during a single, routine blood test. Most recently, we found that very preterm infants who received Calmer treatment for 3 continuous weeks had 25% greater head growth compared to controls. However, we do not know if/how Calmer treatment affects brain development in very preterm infants.

Objectives: We will gather pilot data for a larger trial to examine differences in brain structural and functional development in very preterm infants who receive Calmer treatment for 2-3 consecutive weeks compared to controls.

Methods: 22 infants born 26-30 weeks GA admitted to BC Women's Hospital NICU will be randomized to either control (n=11) or treatment groups (n=11; Calmer for 2-3 continuous weeks, 3 hours/day minimum treatment). Infants from both groups will undergo feed and bundle MRI scans at term-equivalent age using high resolution volumetric, diffusion and resting-state functional MRI to explore group differences in whole-brain volumes and structural and functional connectivity. Images will be processed using existing quantitative neonatal imaging analysis pipelines in the Selvanathan and Weber labs at BC Children's Hospital Research Institute. Analyses will include: measures of trial feasibility and description of brain differences between groups.

Significance: Ultimately, Calmer may support healthy brain maturation optimizing the neurodevelopment of vulnerable infants in Canada and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm infants admitted to the NICU at the BC Women's Hospital

Exclusion Criteria: Infants who have

* Congenital anomalies;
* Born small for GA (per medical admission history);
* History of birthing parent substance use in pregnancy;
* Ongoing infection at the time of enrollment;
* Pre-existing cardiovascular instability defined by shock/hypotension/need for cardiovascular drugs;
* Receiving paralytic drugs;
* Major neurological injury (e.g. hypoxic ischemic encephalopathy, hemorrhage/stroke; VP shunt);
* Beyond the 30th completed week GA (30 weeks + 6 days) at enrollment.

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Brain Volumes | When each participant reaches 40 weeks post-conceptual age and return for their MRI scan
  Anatomical analysis: Anatomical images (T2w) will be manually inspected for quality control. Images with very poor tissue contrast or motion artefacts will be rejected. T2w images will be bias-field corrected using ANTs N4ITK. The images will then be skull-stripped and segmented using the dHCP anatomical pipeline to calculate total and sub-regional brain volumes.
Brain Functional Connectivity | When each participant reaches 40 weeks post-conceptual age
  Resting state fMRI analysis: Fieldmaps will be generated using the dual-echo EPI and magnitude scan. The dHCP functional pipeline will be implemented to achieve distortion-correction and motion-correction, register the functional image to the corresponding T2w structural image, generate a transform matrix from functional space to the 40-week T2w template; and we will perform temporal high-pass filtering (150 s high-pass cutoff) and independent component analysis (ICA) denoising using ICA FIX. Scans with a mean FD > 1 mm will be excluded. The dHCP functional pipeline will then be run on all subjects using the study-specific training file. Spatial smoothing of 5 mm will be applied using FSL's SUSAN and grand mean intensity normalization will be computed. Functional connectivity measures will be computed using the CONN toolbox.
Brain Fractional Anisotropy | When participants reach term-equivalent age
  Diffusion tensor imaging analysis: The dHCP neonatal dMRI data processing pipeline will be used to pre-process the diffusion weighted images. Briefly, opposite phase b0 images are used to estimate the off-resonance field that is then used in the simultaneous correction of motion artefacts, susceptibility-induced and eddy current distortions. Data will then be super-resolved and, after pre-processing is complete, local diffusion and microstructural models are fitted in every voxel and averaged to calculate mean fractional anisotropy.

SECONDARY OUTCOMES:
Clinical weight measures | From the start of study treatment (or enrolment if Control group) to 2-3 weeks later, at the end of intervention exposure.
  Weight: infant weight in kilograms captured when enrolled in the study (i.e. baseline T1) and end of experimental phase (2-3 weeks later; T2)
  We will use the weight measure to determine changes between baseline and the end of treatment.
Head growth measures | From the start of study treatment (or enrolment if Control group) to 2-3 weeks later, at the end of intervention exposure.
  Head circumference: infant head circumference in centimetres (occipito-frontal circumference) captured when enrolled in the study (i.e. baseline T1) and end of experimental phase (2-3 weeks later; T2).
  We will use the head circumference measures to determine changes between baseline and the end of treatment.

OTHER OUTCOMES:
Trial feasibility | 2 years from the start of the study
  Consent rate: overall average consent rate of infants/month
Trial feasibility | 2 years from the start of the study
  Protocol delivery: % of on/off protocol infants
Trial feasibility | 2 years from the start of the study
  Outcome measures: % of infants with complete primary outcome data
Trial feasibility | 2 years from the start of the study
  Rate/nature of safety issues

CONTACTS AND LOCATIONS:
Overall Officials: Manon Ranger, PhD, Principal Investigator — University of British Columbia; Liisa Holsti, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital & Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
As part of this study, participants' de-identified research data may be shared in a public database when the research is published. Sharing this deidentified data helps make research more transparent and allows others to double-check the results. It also means that other researchers can use the data for different studies in the future, beyond the scope of this current study. The exact details have not been decided yet.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: When the research findings are published.
Access Criteria: We have not decided on these details.
URL: https://notcurrentlyavailable.ca

REFERENCES:
- [Result] Holsti L, MacLean K, Oberlander T, Synnes A, Brant R. Calmer: a robot for managing acute pain effectively in preterm infants in the neonatal intensive care unit. Pain Rep. 2019 Mar 14;4(2):e727. doi: 10.1097/PR9.0000000000000727. eCollection 2019 Mar-Apr. PMID 31041426
- [Result] Ranger M, Albert A, MacLean K, Holsti L. Cerebral hemodynamic response to a therapeutic bed for procedural pain management in preterm infants in the NICU: a randomized controlled trial. Pain Rep. 2021 Jan 12;6(1):e890. doi: 10.1097/PR9.0000000000000890. eCollection 2021 Jan-Feb. PMID 33490850